CLINICAL TRIAL: NCT00506038
Title: Phase 2 Study of the Fine Needle Technique on Calcific Tendinitis
Brief Title: Efficacy Study of Fine Needle Technique on Calcific Tendinitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAF01-HMO-CTIL
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2008-11

CONDITIONS: Tendinitis
Keywords: Calcific Tendinitis
MeSH Terms: conditions — Tendinopathy

INTERVENTIONS:
Procedure: fine needle technique

SUMMARY:
Background: Calcific tendinitis of the rotator cuff may cause chronic pain at the shoulder. Sometimes the pain can lead to a serious impairment in the daily life.

One of the most efficient treatments is percutaneous needle aspiration using ultrasound guidance.

This treatment includes identification the tendonitis with US or screening , local anesthesia and then puncturing the calcium in the rotator cuff many times. The treatment is short 5-10 minutes, relatively cheap ,safe and usually with good outcomes. However in the literature there is a lack of controlled prospective trials.

Our goal is to set a study that will evaluate this treatment between two groups:

1. Puncturing the calcium in the rotator cuff 15 times (the experiment group)
2. Puncturing the calcium in the rotator cuff twice (the controlled group)

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above.
2. 6 months of pain in the shoulder.
3. Positive IMPING and sensitivity on SST.
4. Calcification above 1 cm in one of the dimensions by US or aray of the shoulder.
5. Completed conservative treatment: physiotherapy or analgesics.

Exclusion Criteria:

1. Diabetes, Nephrological diseases
2. RC tear according to US.
3. Prior operation in this shoulder
4. Steroids injection in the last three months.
5. A patient that is in the absorption phase of the tendinitis
6. Pregnancy
7. Coagulation System impairments

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ori Safran, MD, Principal Investigator — Hadassah Medical Organization; Charles Milgrom, Prof., Study Chair — Hadassah Medical Organization